CLINICAL TRIAL: NCT05190692
Title: A Prospective Study of the Benefits of Simulators in Improving Obstetric Vaginal Examination Skills
Brief Title: Role of Simulators in Improving Obstetric Vaginal Examination Skills
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Lecturer of Obstetrics and Gynecoloy department, Cairo University
Other Study IDs: Simulators in obstetrics
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Labour
Keywords: Simulator_vaginal examination_labour

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Use simulators in Obstetrics vaginal examination — Two simulators will be used in the study:
  (1st ) : PROMPT Flex Birthing Simulator Advanced - Light (PRODUCT NO. 80106).UK, 2020 .
  2nd): PROMPT Flex Cervical Dilatation & Effacement Module -Light (PRODUCT NO. 80102),Uk,2020.
  Both will be used to perform obstetric vaginal examination before examination of patients

SUMMARY:
A prospective study will be performed at the Department of Obstetrics and Gynecology at (VESSALKA unit),at El kasr Al_Ainy hospital, cairo university. Sample of house officers without obstetric experience in vaginal examination that will begin their clinical rotation in the department will be eligible for inclusion in the study. All patients involved in the study must not be high risk pregnancy nor have any indication of cesarean section and they will be examined by house officers in the first stage of labor. House officers and patients will provide verbal informed consent for participation in the study .all house officers assigned in the obstetric and gynecology department for their clinical rotation at the time of study will receive about a (30-mins) standardized course summarizing how to perform an obstetric vaginal examination . All house officers assigned in the study will be trained on vaginal examination simulators in about (15) training sessions and giving them a score to each one about their performing results on simulators.

DETAILED DESCRIPTION:
This prospective study will be done on a group of house officers without obstetric experience in vaginal examination.

They will perform multiple vaginal examination training procedures using a simulators in about (15) training sessions and giving them a score to each one then testing them on patients who are in the 1st stage of labor and giving them another score after collection of their results .

All house officers will report the findings of examinations of each time in terms of six items (1): cervical dilatation. (2): cervical effacement. (3): presenting part and position. (4): caput or not. (5): station. (6): condition of membrane intact or ruptured.

The findings that will be obtained by the house officers will then be revised by the same staff experienced obstetrician and gynaecologist {whose answers will be considered to be the gold standard} who will examine the same patients at the same time for accuracy of results.

Two simulators will be used in the study:

1. st ) : PROMPT Flex Birthing Simulator Advanced - Light (PRODUCT NO. 80106).UK, 2020 .
2. nd) : PROMPT Flex Cervical Dilatation & Effacement Module -Light (PRODUCT NO. 80102),Uk,2020

ELIGIBILITY:
Inclusion Criteria:

* House officers must be without any experience in vaginal examination at the start of study.
* Study group must attend at least (15) simulator training sessions before testing them.

Exclusion Criteria:

* House officers with any experience in vaginal examination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - House officers must be without any experience in vaginal examination at the start of study.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
learning curve and efficiency of vaginal examination interpretation. Learning curve and efficiency of vaginal examination interpretation. | Five months
  Simulation training on non experienced house officers will improving or not their vaginal examination skills before performing it on real pregnant women in labor

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Kasr Alainy hospital-cairo University, Cairo
  - Obstetrics and gynecology department at kasralainy hospital, Cairo
  - Cairo University, Giza

IPD SHARING:
Plan to Share IPD: Undecided
Should vaginal examination simulator be included in the training curriculum for each house officers during their clinical rotation in gynecology and obstetric department?